CLINICAL TRIAL: NCT00663468
Title: Treatment of Sub-capital Fractures of Hip Joint by Using TriboFit™ Acetabular Buffer
Status: Terminated | Type: Observational
Why Stopped: Lead surgeon retired.
Sponsor: Active Implants (Industry)
Responsible Party: Sponsor
Other Study IDs: TLV-0021-08
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Hip Fractures
Keywords: determine changes in patient pain level; determine changes in patient functionality; determine changes in patient life quality
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A

SUMMARY:
The purpose of this study is to determine the performance and efficacy during 6 and 12 month post operation.

1. determine changes in patient pain level
2. determine changes in patient functionality
3. determine changes in patient life quality

ELIGIBILITY:
Inclusion Criteria:

* Female or male that is not younger than 60 years old.
* Patient suffers from hip fracture that will need hip arthroplasty.
* Patient that weight less than 150Kg
* Patient femur head diameter between 40mm - 50mm
* Mentally normal
* Patient that could walk before suffering from hip fracture
* Patient that willing to cooperate with the doctor
* Patient that signed on the acceptance form

Exclusion Criteria:

* Patient that does not willing to cooperate with the doctor
* Patient that is legally rejected
* Patient that suffer from cancer
* Patient that had passed amputation in is limbs
* Patient that is paralysis
* Patient that passed CVA or TIA
* Patient that still recovering from hard wounds or surgery
* Patient that suffer from infection in the hip joint

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09-16 (Actual); Study Completion 2009-09-16 (Actual)